CLINICAL TRIAL: NCT06359886
Title: B-lynch Transverse Compression Suture in the Prophylaxis and Control of Postpartum Heamorrhage in Patients With Placenta Previa: A Pilot Study
Brief Title: B-lynch Transverse Compression Suture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Zeerban, Doctor, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FMASU MD 292/2022
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Intervention Model Description: A Pilot Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B-Lynch Transverse Compression Suture (Experimental): Transverse B-Lynch suture will be performed to these patients as a method of controlling postpartum heamorrhage in placenta previa patients
  Interventions: Procedure: B-Lynch Transverse Compression Suture

INTERVENTIONS:
Procedure: B-Lynch Transverse Compression Suture — closure of uterine and utero ovarian arteries bilaterally with one suture
  Other Names: B-Lynch Transverse Compression Suture using 1 Polyglactin 910 with a 70mm ½ circle needle mounted on a 90 cms suture

SUMMARY:
Is B-Lynch transverse compression suture safe and effective in controlling excessive blood loss during conservative management of women with placenta previa?

DETAILED DESCRIPTION:
To perform B-Lynch Transverse Compression Suture the investigators will use the suture material 1 Polyglactin 910 with a 70mm ½ circle needle mounted on a 90 cms suture. the investigators will use the needle blunt ended to puncture the uterus 3 cms above the upper margin of the incision posteriorly and behind the vascular bundle.

The needle is retrieved through the cavity of the uterus and pulled inferiorly with the suture material lying on the posterior wall of the uterine cavity. The needle then perforates the posterior wall of the uterus 1-3 cms below the inferior margin of the Caesarean incision and exists behind the vascular bundle of the same side of the uterus retrieved and runs on the surface of the lower segment below the incision margin parallel to it and taking a 1 cm bite of tissue for stabilization running to the other side.

After encircling the para-uterine vasculature, the needle then perforates the posterior side of the uterus behind the vascular bundle entering the uterine cavity 1-3 cm below the inferior margin of the Caesarean incision. The suture can lie freely on the posterior wall of the uterine cavity and exists 3 cms above the upper margin of the Caesarean incision. It exits posteriorly and behind the vascular bundle to meet the suture from the other side.

It is essential that the ureters are identified by palpation or visual observation after the bladder is displaced inferiorly and held by traction. Any observed bleeding should be dealt with in the usual way. At the end of the suture application and before tying the knots, the lower segment is compressed again transversely whilst the suture is held taut to ensure that bleeding has ceased by swabbing the vagina again.

A wide pore drain will be inserted in the Douglas pouch, and the abdominal wall will be repaired.

ELIGIBILITY:
Inclusion Criteria:

1. Single gestation
2. Elective CS for placenta preiva (diagnosed by transvaginal ultrasound).
3. Muliparity (para 2 or more).

Exclusion Criteria:

1. Morbidly adherent placenta: accrete, increta or percreta, diagnosed by abdominal and/or transvaginal ultrasound.

   • Ultrasonographic features of morbidly adherent placentas:
   * Loss of Retro-placental sonolucent zone.
   * Vascular lacunae.
   * Myometrial thinning.
   * Interruption of the bladder border.
2. More than 3 previous C.S.
3. Severely haemodynamic instablility needing immediate hysterectomy.
4. Patients with the cardiac, hepatic, renal or thromboembolic disease
5. Patients with coagulopathy:

   * Receiving anticoagulant therapy.
   * With thrombocytopenia or thrombasthenia.
   * Known coagulation factor defect.
6. Distorted uterus as unicornuate, bicornuate, fibroid uterus and adenomyosis uteri.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females with Placenta Previa
Enrollment: 25 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | 2 days following the procedure
  Number of towels and blood in suction reservoir
Postoperative blood loss | 2 days following the procedure
  Postoperative blood loss in the drain bag
Number of received blood components | 2 days following the procedure
  Packed RBC's
Peripartum haemoglobin level drop | 2 days following the procedure
  Difference between pre and postoperative hemoglobin level

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Statistical data discussion conclusion
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Avilable from now onward
Access Criteria: Transverse B-Lynch Placenta previa